CLINICAL TRIAL: NCT05499832
Title: Safety and Efficacy of Intra-arterial Tenecteplase for Noncomplete Reperfusion of Intracranial Occlusions
Acronym: TECNO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-00388
Record Dates: First submitted 2022-04-26; First posted 2022-08-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Medical Treatment (standard of care) (No Intervention): Patients will receive standard of care as per current ESO guidelines.
- Intra-arterial Tenecteplase (Experimental): Patients will receive intra-arterial administration of Tenecteplase using a standard approved microcatheter.
  Interventions: Drug: Tenecteplase

INTERVENTIONS:
Drug: Tenecteplase — Patients randomized to IA treatment will receive IA TNK via a standard approved microcatheter positioned as close as possible to the residual occlusion site or as distal as possible in the originating vessel if multiple residual occlusions exists.
  Arms: Intra-arterial Tenecteplase

SUMMARY:
TECNO is a multicenter, prospective, randomized, open label, blinded endpoint (PROBE) proof-of-concept trial evaluating if additional administration of intra-arterial Tenecteplase (TNK) improves reperfusion in patients with incomplete mechanical thrombectomy (MT). For this purpose, 156 adult participants experiencing an acute ischemic stroke due to a large vessel occlusion with incomplete reperfusion with residual occlusions after MT will be randomly assigned to receive 3mg intra-arterial (IA) TNK or best medical treatment. Recruitment will occur at 20 academic tertiary stroke care centers in Switzerland, Spain, Belgium, and Germany and patients are followed up for 90 days after the index event. Showing superiority for reperfusion outcomes would have a major impact on the future management of stroke patients.

ELIGIBILITY:
Inclusion Criteria

* Informed consent
* Age ≥18 years
* Clinical signs consistent with an acute ischemic stroke
* Patient had an initial vessel occlusion in the anterior or posterior circulation defined as intracranial ICA, M1, M2, M3, A1, A2, P1 or P2
* Patient has undergone endovascular stroke treatment
* Onset to randomization no later than < 705 minutes (11h 45min) after symptom-onset/last-seen well.
* Incomplete reperfusion defined as any of the following:

  1. For ICA/M1: TICI2b/2c (50-99%) reperfusion after endovascular treatment without mechanically amendable target-occlusion (as per definition by the interventionalist).
  2. For A1/A2, P1/P2, M2/M3: TICI2a/2b/2c (1-99%) reperfusion after endovascular treatment without mechanically amendable target-occlusion (as per definition by the interventionalist).
  3. Any emboli to new territory without mechanically amendable target-occlusion (as per definition by the interventionalist).
* Signs of early ischemic changes of non-contrast CT Alberta Stroke Program Early CT Score (ASPECTS) ≥5 (for DWI-ASPECTS ≥ 4, for DWI-ASECTS: a region must have diffusion abnormality in 20% or more of its volume to be considered DWI-ASPECTS positive)

Exclusion Criteria

* Acute intracranial hemorrhage
* Contraindication to MRI (e.g. pacemaker)
* Any severe bleeding within the past 6 months, which would prevent administration of intravenous thrombolysis in clinical routine Major surgery in the past 2 months with severe risk of bleeding, which would prevent administration of intravenous thrombolysis in clinical routine
* Intake of Vitamin K antagonists with INR >1.7
* Platelets < 50,000
* Non-controlled hypertension (defined as SBP >185 mmHg or DBP >110 mmHg refractory to treatment)
* Active dyspeptic ulcer
* Known arterial aneurysm
* Known neoplasms with risk of bleeding
* Severe liver fibrosis or portal hypertension
* Acute pericarditis
* Acute endocarditis
* Acute pancreatitis
* Known allergy to TNK or Gentamicin or other additives/auxiliaries (Polysorbatum 20, L-Argininum, Acidum phosphoricum)
* Known Renal failure either as defined by a serum creatinine > 3.0 mg/dl (or 265.2 μmol/l) or glomerular Filtration Rate [GFR] < 30 or as subject who required hemodialysis/peritoneal dialysis
* Radiological confirmed evidence of mass effect or intracranial tumor (except small meningioma)
* Radiological confirmed evidence of cerebral vasculitis
* Calcified thrombi
* Pregnancy or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Early reperfusion of the residual intracranial occlusion(s) | 25 minutes after randomization
  Defined by reperfusion improvement on angiography images
Late reperfusion of the residual intracranial occlusion(s) | 24 hours ±6 hours
  Defined by complete reperfusion on perfusion imaging

SECONDARY OUTCOMES:
Degree of disability or dependence assessed by the modified ranking scale (mRS) (shift analysis) | 90 days+/-15 days
  mRS
Normalized change in National Institute of Health Score Scale (NIHSS) | 24 hours +/- 6 hours post-randomization
  NIHSS
Change in National Institute of Health Score Scale (NIHSS) | 90 days +/- 15 days post-randomization
  NIHSS
Quality of life as assessed by the EuroQol 5D-3L (EQ-5D-3L) | 90 days +/- 15 days
  EuroQol 5D-3L
All-cause mortality | 90 days
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Urs Fischer, PhD, Study Director — NCTU
Locations (51):
- Austria (4):
  - LKH-Universitätsklinikum Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Kepler Universitätsklinikum GmbH, Linz
  - Christian-Doppler-Klinik Salzburg, Salzburg
- Belgium (7):
  - Hôpital universitaires de Bruxelles, Anderlecht
  - AZ Sint Jan Brugge AV, Bruges
  - UZ Brussel, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Gasthuisberg Leuven, Leuven
  - Clinique CHC MontLégia, Liège
- University Hospital Helsinki, Helsinki, Finland
- Germany (20):
  - Universitätsklinikum Augsburg, Augsburg
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Bremen-Mitte, Bremen
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Halle (Saale), Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Universitätsklinikum Magdeburg A. ö. R., Magdeburg
  - Universitätsmedizin Mannheim, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum der Universität München, München
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Universitätsklinikum Münster, Münster
  - Städtisches Klinikum Sollingen, Solingen
  - Universitätsklinikum Tübingen, Tübingen
- Netherlands (2):
  - Amsterdam UMC, Amsterdam
  - Leiden UMC, Leiden
- Portugal (5):
  - Hospital de Braga, Braga
  - Hospital Nelio Mendonca Funchal, Funchal
  - Lisbon Central University Hospital, Lisbon
  - Hospital Eagas Moniz, Lisbon
  - Hospital Santo Antonio, Porto
- Switzerland (12):
  - Kantonsspital Aarau AG, Aarau
  - Kantonsspital Aarau, Aarau
  - Universitätsspital Basel, Basel
  - Universitätsspital Bern, Bern
  - Hôpitaux universitaires de Genève, Geneva
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - University Hospital of Lausanne, Lausanne
  - Kantonsspital Luzern, Lucerne
  - Ospedale Regionale di Lugano, Lugano
  - Kantonsspital St.Gallen, Sankt Gallen
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mujanovic A, Windecker D, Cimflova P, Meinel TR, Seiffge DJ, Auer E, Boulouis G, Arnold M, Serrallach BL, Rohner R, Janot K, Dobrocky T, Hill MD, Goyal M, Piechowiak EI, Gralla J, Fischer U, Kaesmacher J. Natural Evolution of Incomplete Reperfusion in Patients Following Endovascular Therapy After Ischemic Stroke. Stroke. 2025 Feb;56(2):447-455. doi: 10.1161/STROKEAHA.124.049641. Epub 2024 Nov 20. PMID 39567366